CLINICAL TRIAL: NCT05396118
Title: Phase IIa Clinical Trial: Feasibility Study on Non-Invasive Simultaneous Hyperpolarized [1-13C]Pyruvate Magnetic Resonance Spectroscopy and 18F-FDG PET (hyperPET) for Metabolic Imaging in Patients With Cancer
Brief Title: Simultaneous Hyperpolarized [1-13C]Pyruvate and 18F-FDG PET/MRS in Cancer Patients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mathias Loft, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK_2021_HP
Record Dates: First submitted 2022-05-12; First posted 2022-05-31 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Neuroendocrine Tumors; Neuroendocrine Carcinoma; Neuroendocrine Carcinoma Metastatic; Lymphoma; Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Neuroendocrine Tumors; Carcinoma, Neuroendocrine; Lymphoma; Sarcoma | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Injection of 18F-FDG and injections of hyperpolarized [1-13C]Pyruvate and subsequent PET/MRI/MRS scan
  Interventions: Drug: 18F-FDG; Drug: Injection of hyperpolarized [1-13C]Pyruvate; Procedure: PET/MR/MRS/MRSI scanning

INTERVENTIONS:
Drug: 18F-FDG — Injection of 4 MBq/kg of 18F-FDG followed by dynamic positron emission tomography (PET) imaging
  Other Names: 18F-fluorodeoxyglucose; fluorodeoxyglucose-F-18; [18F]F-FDG
Drug: Injection of hyperpolarized [1-13C]Pyruvate — Injection of one bolus of 0.43 ml/kg of approximately 250 mM hyperpolarized [1-13C]Pyruvate followed by magnetic resonance spectroscopy (MRS) / magnetic resonance spectroscopy imaging (MRSI). After a 5-30 min pause, injection of a second bolus of 0.43 ml/kg of approximately 250 mM hyperpolarized [1-13C]Pyruvate followed by MRS / MRSI.
Procedure: PET/MR/MRS/MRSI scanning — Regional dynamic PET acquisition for up to 90 minutes following 18F-FDG injection is performed focused on a region-of-interest (ROI). Anatomical magnetic resonance imaging (MRI) is performed in the ROI, including diffusion weighted imaging (DWI) and contrast enhanced imaging (DCE). MRS/MRSI is performed following the injections of hyperpolarized [1-13C]Pyruvate.

SUMMARY:
Prospective phase 2a clinical trial to demonstrate proof-of-concept for simultaneous hyperpolarized [1-13C]pyruvate and 18F-FDG for positron emission tomography (PET) and MRS (magnetic resonance spectroscopy) in a PET/MR scanner in patients with cancer.

DETAILED DESCRIPTION:
PET imaging with 18F-FDG is a well established method for non invasively assessing the intracellular glucose accumulation. 18F-FDG PET is used in many applications with diagnosing and staging of patients with cancer being one of the primary indications. Once internalized into the cell, 18F-FDG is phosphorylated to the metabolically inactive 18F-FDG-6-phosphate. Therefore it is not possible to determine what happens to the downstream glucose metabolites. In particular, it is not possible to determine the conversion into lactate, which is upregulated in many cancers. The upregulation of lactate conversion in cancers, even in presence of oxygen, is known as the Warburg effect.

Hyperpolarized [1-13C]pyruvate MRS makes is possible to circumvent this limitation. The technique makes is it possible to follow the downstream fate of the glycolysis intermediate, pyruvate, and in particular makes is is possible to non-invasively and in in real time measure the glycolytic conversion of pyruvate into lactate as a direct measure of the Warburg effect.

When using a PET/MR scanner, it is possible to simultaneous measure the glucose influx with 18F-FDG and the conversion of pyruvate into lactate with hyperpolarized [1-13C]pyruvate. In this way, the two modalities provide complementary information on the in vivo glycose metabolism.

The prospective phase 2a project will include up to 15 patients diagnosed with breast cancer, gastro-entero-pancreatic neuroendocrine neoplasms (GEP-NEN) of all grades (G1, G2, G3)., lymphomas or sarcomas The aim is to demonstrate proof-of-concept for the feasibility of simultaneous acquisition of hyperpolarized [1-13C]pyruvate MRS and 18F-FDG PET imaging in a PET/MR scanner in cancer patients to allow for simultaneous measurements of overall tumor pyruvate-to-lactate conversion parameters on MRS and glucose influx with 18F-FDG on PET.

Included patients are injected with a standard dose of radioactive 18F-FDG. Subsequent dynamic PET acquisition is performed for up to 90 minutes after injection on an area-of-interest covering pre-specified tumor lesion(s). Regional anatomical magnetic resonance imaging (MRI) is performed, including diffusion weighted imaging (DWI) and contrast enhanced imaging (DCE). MRS/MRSI is performed following the injection(s) of hyperpolarized [1-13C]Pyruvate.

When available, resected tumor tissues samples from surgical specimens or biopsies obtained in relation to routine clinical procedures will be collected and analyses of enzymes and markers of glycolytic metabolism will be performed ex vivo and compared with the in vivo data from PET/MRS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer, gastro-entero-pancreatic neuroendocrine neoplasms (GEP-NEN) grades G1, G2 or G3, lymphoma or sarcoma
* Measurable solid tumor of at least 1.5 cm
* Capable of understanding the patient information in Danish and giving full informed consent

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Weighs above 140 kg and/or with abdominal circumference exceeding the gantry of the PET/MR coil (120 cm)
* History of allergic reaction attributable to compounds of similar chemical or biologic composition to 18F-FDG or pyruvate
* Patients who are unable to lie in the MR scanner for up to 90 minutes
* Pace-maker
* Metallic implantations within the past 6 weeks
* Non-MR compatible implants
* Claustrophobia
* Participants who have not fasted for a minimum of 4 hours prior to the planned scan time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Whole-tumor lactate/pyruvate ratio measured with MRS | Up to 10 minutes after injection of hyperpolarized [1-13C]Pyruvate
  Whole-tumor lactate/pyruvate ratio measured with MRS in regions-of-interest covering the tumor lesion(s) following injection of hyperpolarized [1-13C]Pyruvate
Whole-tumor glucose uptake measured with PET (static) | Approximately 60 minutes after injection of 18F-FDG
  Whole-tumor standardized uptake values (SUV): SUVmean and SUVmax measured with PET in regions-of-interest covering the tumor lesion(s) approximately 60 minutes after injection of 18F-FDG
Whole-tumor glucose uptake measured with PET (dynamic) | Up to 90 minutes after injection of 18F-FDG
  Whole-tumor glucose influx rate constant (Ki) derived from dynamic PET in regions-of-interest covering the tumor lesion(s) following injection of 18F-FDG
Correlation between whole-tumor lactate/pyruvate ratio measured with MRS and tumor glucose uptake measured with PET (static) | Approximately 60 minutes after injection of 18F-FDG
  Correlation between whole-tumor lactate/pyruvate ratio measured with MRS and whole-tumor SUVmean and SUVmax measured with PET in regions-of-interest covering the tumor lesion(s)
Correlation between whole-tumor lactate/pyruvate ratio measured with MRS and tumor glucose uptake measured with PET (dynamic) | Up to 90 minutes after injection of 18F-FDG
  Correlation between whole-tumor lactate/pyruvate ratio measured with MRS and whole-tumor Ki measured with PET in regions-of-interest covering the tumor lesion(s)

SECONDARY OUTCOMES:
Correlation between measurements of in vivo glycolytic markers based on PET/MRS and enzymes involved in glycolytic metabolism based on ex vivo analyses | Up to 90 minutes after injection of 18F-FDG
  Ex vivo measurements of enzymes, regulatory proteins and transporters involved in glucose and pyruvate/lactate transcellular transport and in glycolysis on resected matched tumor tissue samples (if available) and the correlation with the primary endpoints (whole-tumor lactate/pyruvate ratio, SUVmax, SUVmean, and Ki)

OTHER OUTCOMES:
Tertiary (exploratory) Outcome Measure: Spatially mapped tumor lactate/pyruvate ratios measured with MRS | Up to 10 minutes after injection of hyperpolarized [1-13C]Pyruvate
  Spatially mapped tumor lactate/pyruvate ratios measured with MRS in segmented regions-of-interest within the tumor lesion(s) following injection of hyperpolarized [1-13C]Pyruvate
Tertiary (exploratory) Outcome Measure: Spatially mapped tumor glucose uptakes measured with PET (static) | Approximately 60 minutes after injection of 18F-FDG
  Spatially mapped SUVmean and SUVmax measured with PET in segmented regions-of-interest within the tumor lesion(s) approximately 60 minutes after injection of 18F-FDG
Tertiary (exploratory) Outcome Measure: Spatially mapped tumor glucose uptakes measured with PET (dynamic) | Up to 90 minutes after injection of 18F-FDG
  Spatially mapped glucose influx rate constants (Ki) derived from dynamic PET in segmented regions-of-interest within the tumor lesion(s) following injection of 18F-FDG
Tertiary (exploratory) Outcome Measure: Correlation between spatially mapped lactate/pyruvate ratios measured with MRS and tumor glucose uptakes measured with PET (static) | Approximately 60 minutes after injection of 18F-FDG
  Correlation between spatially mapped tumor lactate/pyruvate ratios measured with MRS and spatially mapped SUVmean and SUVmax measured with PET in segmented regions-of-interest within the tumor lesion(s)
Tertiary (exploratory) Outcome Measure: Correlation between spatially mapped lactate/pyruvate ratios measured with MRS and tumor glucose uptakes measured with PET (dynamic) | Up to 90 minutes after injection of 18F-FDG
  Correlation between spatially mapped tumor lactate/pyruvate ratios measured with MRS and spatially mapped glucose influx rate constants (Ki) derived from dynamic PET in segmented regions-of-interest within the tumor lesion(s)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Loft, MD, Principal Investigator — Rigshospitalet, Denmark; Andreas Kjaer, MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not publicly available due to protection of personal data according to data protection regulations and medical confidentiality.